CLINICAL TRIAL: NCT03275740
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO -CONTROLLED, FIRST-IN-HUMAN TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF PF 06755347 AFTER SINGLE ASCENDING INTRAVENOUS AND SUBCUTANEOUS DOSING IN HEALTHY ADULT MALE PARTICIPANTS AND OPEN-LABEL AFTER SINGLE SUBCUTANEOUS DOSING IN MALE AND FEMALE PARTICIPANTS WITH PERSISTENT OR CHRONIC PRIMARY IMMUNE THROMBOCYTOPENIA
Brief Title: A First in HumanTrial to Evaluate The Safety, Tolerability, And Pharmacokinetics Of PF-06755347
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor has decided to terminate the above referenced clinical study for business reasons. There were no safety concerns that led to this decision and there was no impact to participant safety.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: B7801001; 2018-003315-21 (EudraCT Number)
Record Dates: First submitted 2017-07-06; First posted 2017-09-08 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Primary Immune Thrombocytopenia; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Intervention Model Description: single ascending dose study
Who Masked: Participant, Investigator
Masking Description: Double blind (investigator and subject), sponsor open in healthy male participants. Masking will not be applied for participants with ITP (all ITP participants will receive PF-06755347).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PF-06755347 intravenous healthy participant (Experimental): intravenous administration
  Interventions: Drug: PF-06755347 intravenous healthy participant
- Placebo intravenous healthy participant (Placebo Comparator): intravenous administration
  Interventions: Drug: Placebo intravenous healthy participant
- PF-06755347 subcutaneous healthy participant (Experimental): subcutaneous administration
  Interventions: Drug: PF-06755347 subcutaneous healthy participant
- Placebo subcutaneous healthy participant (Placebo Comparator): subcutaneous administration
  Interventions: Drug: Placebo subcutaneous healthy participant
- PF-06755347 subcutaneous ITP (Experimental): subcutaneous
  Interventions: Drug: PF-06755347 subcutaneous ITP

INTERVENTIONS:
Drug: PF-06755347 intravenous healthy participant — Single doses of PF-06755347 will be administered intravenously dose levels 1, 2, 3, 4, 5, and 6.
  Arms: PF-06755347 intravenous healthy participant
Drug: Placebo intravenous healthy participant — Placebo comparator
  Arms: Placebo intravenous healthy participant
Drug: PF-06755347 subcutaneous healthy participant — single doses of PF-06755347 will be administered subcutaneously at dose levels of SC1, SC2, SC3, SC4, and SC5.
  Arms: PF-06755347 subcutaneous healthy participant
Drug: Placebo subcutaneous healthy participant — placebo comparator
  Arms: Placebo subcutaneous healthy participant
Drug: PF-06755347 subcutaneous ITP — single doses of PF-06755347 will be administered subcutaneously at 2 dose levels tested in healthy participants
  Arms: PF-06755347 subcutaneous ITP

SUMMARY:
This phase 1 single ascending dose study will provide a first in human assessment of safety and tolerability of PF-06755347 in healthy adult males as well as adult males and females with Immune Thrombocytopenia (ITP). Pharmacokinetics and pharmacodynamics will also be evaluated.

ELIGIBILITY:
Inclusion Criteria Healthy male participants:

* at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including oral temperature, blood pressure (BP) and pulse rate measurement, pulse oximetry, 12 lead ECG or clinical laboratory tests.
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Chest X ray with no evidence of current, active tuberculosis (TB) or previous inactive TB, general infections, heart failure, malignancy, or other clinically significant abnormalities taken at Screening or within 3 months prior to Screening and read by a qualified radiologist.

Exclusion Criteria for Healthy male participants:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Participants with a history of autoimmune disorders and other conditions that compromise or impair the immune system (including but not limited to: Crohns Disease, rheumatoid arthritis, scleroderma, systemic lupus erythematosus, Graves disease, and asthma) or have a current positive result for the following; rheumatoid factor, anti-nuclear antibody, or abnormal free triiodothyronine (T3), free thyroxine (T4), thyroid stimulating hormone (TSH), or thyroid stimulating antibody (TSAb) suggestive of thyroid disease.
* Subjects with a history of allergic or anaphylactic reaction to any drug including immunoglobulin.
* History of active infections within 28 days prior to the screening visit.
* Subjects with a history of or current positive results for any of the following serological tests: Hepatitis B surface antigen (HepBsAg), Hepatitis B core antibody (HepBcAb), Hepatitis C antibody (HCVAb) or human immunodeficiency virus (HIV).
* Subjects with a history of thromboembolic events.
* History of TB or active, latent or inadequately treated TB infection. All positive TB test result(s) are exclusionary
* Male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study.
* Inclusion Criteria for ITP participants:

Female participants may be of childbearing potential or non-childbearing potential.

-Diagnosis of Primary ITP. ITP must be diagnosed in accordance with established guidelines. ITP duration-Persistent (>3 months and ≤12 months) OR Chronic (>12 months).

AND

* Platelet count 30-75 x 10E9/L (inclusive) with criteria achieved on 2 qualifying counts at least 5 days apart and within approx. 10 days of dosing
* Participants must have received and responded to IVIg or corticosteroids as treatment for ITP (response is defined as achievement of platelet count >50 x 109/L and doubling of platelet count from baseline).

  --Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* BMI of 17.5 to 30.5 kg/m2 and a total body weight >40 kg (88 lbs).

Exclusion Criteria for ITP participants

* History of clinically significant hematological (other than ITP), renal, endocrine, metabolic, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Chest X-ray with evidence of current, active TB, previous inactive TB, general infections, heart failure, malignancy, or other clinically significant abnormalities.

Chest x-ray must be taken at Screening or within 3 months prior to Screening and read by a qualified radiologist.

* Any bleeding event requiring medical evaluation or treatment in the 4 weeks prior to screening or current bleeding event that requires treatment.
* Scheduled or anticipated invasive procedures (eg, surgery, dental procedures) within 28 days following PF-06755347 dosing.
* Splenectomy within ≤180 days prior to PF-06755347 dosing or splenectomy planned during the period of the study.
* History of any active autoimmune disorder (other than ITP) or other conditions that may compromise or impair the immune system (including but not limited to: Crohn's Disease, rheumatoid arthritis, scleroderma, systemic lupus erythematosus, Graves' disease, and asthma).
* History of allergic or anaphylactic reaction to any drug including immunoglobulin.
* History of active infections within 28 days prior to the screening visit.
* History of Hepatitis B, Hepatitis C or HIV or current positive results for any of the following serological tests - HBsAg, HBcAb, HCVAb or HIV.
* History of thromboembolic events
* Hemoglobin <9 g/dL.
* Positive Direct Coombs test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States
- Pfizer Clinical Research Unit, Brussels, Belgium
- NZCR (New Zealand Clinical Research) OPCO Limited, Christchurch, New Zealand
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Hammersmith Medicines Research (HMR), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7801001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study planned 14 cohorts, however, it was terminated due to non-safety reasons during Cohort 11, with no further enrollment. Included in this study were all healthy participants, who were randomized to either receive PF-06755347 or placebo by intravenous (IV) or subcutaneous (SC) administration in a 3:1 allocation ratio. A total of 58 participants were dosed in this study: 42 received PF-06755347 and 16 received placebo.
Groups:
- Cohort 1: PF-06755347 0.01 mg/kg IV: Healthy participants received single dose of PF-06755347 0.01 mg/kg IV on Day 1.
- Cohort 2: PF-06755347 0.03 mg/kg IV: Healthy participants received single dose of PF-06755347 0.03 mg/kg IV on Day 1.
- Cohort 3: PF-06755347 0.1 mg/kg IV: Healthy participants received single dose of PF-06755347 0.1 mg/kg IV on Day 1.
- Cohort 4: PF-06755347 0.3 mg/kg IV: Healthy participants received single dose of PF-06755347 0.3 mg/kg IV on Day 1.
- Cohort 5: PF-06755347 1 mg/kg IV: Healthy participants received single dose of PF-06755347 1 mg/kg IV on Day 1.
- Cohort 6: PF-06755347 0.7 mg/kg IV: Healthy participants received single dose of PF-06755347 0.7 mg/kg IV on Day 1.
- Cohort 7: PF-06755347 25 mg SC: Healthy participants received single dose of PF-06755347 25 mg SC on Day 1.
- Cohort 8: PF-06755347 50 mg SC: Healthy participants received single dose of PF-06755347 50 mg SC on Day 1.
- Cohort 9: PF-06755347 100 mg SC: Healthy participants received single dose of PF-06755347 100 mg SC on Day 1.
- Cohort 10: PF-06755347 200 mg SC: Healthy participants received single dose of PF-06755347 200 mg SC on Day 1.
- Cohort 11: PF-06755347 300 mg SC: Healthy participants received single dose of PF-06755347 300 mg SC on Day 1.
- Placebo: Healthy participants received single dose of placebo matching PF-06755347 IV or SC cohorts on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16
Completed | 3 | 3 | 3 | 3 | 2 | 2 | 3 | 6 | 5 | 5 | 3 | 16
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — due to coronaviras disease 2019 (COVID-19) pandemic | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16 | 58
Age, Customized [Count of Participants; unit: Participants]
  18-25 years | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 4 | 15
  26-35 years | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 2 | 3 | 5 | 17
  36-45 years | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 2 | 14
  46-55 years | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 0 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 5 | 6 | 4 | 3 | 16 | 54
  Race: Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Race: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 5 | 5 | 6 | 3 | 14 | 52
  Ethnicity: Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-causality Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, Treatment-related TEAEs, and Discontinuations From Study Due to TEAEs
Description: Adverse event (AE) was any untoward medical occurrence in the participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Serious AE was any untoward medical occurrence that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect, or was considered to be an important medical event. Any events occurring following start of treatment or increasing in severity were counted as treatment-emergent. AEs included both serious and non-serious AEs.
Time Frame: Baseline (Study Day -2) through study completion (Study Day 36 for IV treatment cohorts, and Study Day 71 SC treatment cohorts).
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16
Participants
  All-causality TEAEs | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 3 | 10
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related TEAEs | 2 | 2 | 2 | 2 | 3 | 3 | 2 | 5 | 6 | 4 | 3 | 7
  Discontinuations from study due to TEAEs | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory test included: hematology (hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count, white blood cell count, absolute and percent total neutrophils, eosinophils, monocytes, basophils and lymphocytes),chemistry (blood urea nitrogen/urea and creatinine, fasting glucose, calcium, sodium, potassium, chloride, total carbon dioxide, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin and total protein),urinalysis(pH, qualitative glucose, qualitative protein, qualitative blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, microscopy, urinary albumin to creatinine ratio and urinary protein to creatinine ratio) and other tests. Abnormality was determined by the investigator. Only lab abnormalities with at least 1 occurrence in participants are reported.
Time Frame: Baseline, Study Days 1, 2, 4, 6, 8, 11, 15, 22, 29 and 36 for IV treatment cohorts, and Baseline, Study Days 1, 2, 3, 4, 6, 8, 11, 15, 22, 29, 36, 50 and 71 for SC treatment cohorts.
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Healthy subjects received single dose of placebo matching PF-06755347 IV or SC cohorts on Day 1.
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16
Participants
  Mean Platelet Volume > 1.1 x upper limit of normal (ULN) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
  Ery. Mean Corpuscular Volume <0.9 x lower limit of normal (LLN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Leukocytes <0.6 x LLN | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes <0.8 x LLN | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1
  Ery. Mean Corpuscular Hemoglobin < 0.9 x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphocytes/ Leukocytes >1.2 x ULN: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 1 | 2 | 5 | 1 | 11
  Lymphocytes/ Leukocytes >1.2 x ULN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils <0.8 x LLN | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
  Neutrophils >1.2 x ULN | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils >1.2 x ULN | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
  Eosinophils/Leukocytes >1.2 x ULN: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 1 | 2 | 5 | 1 | 11
  Eosinophils/Leukocytes >1.2 x ULN | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
  Monocytes >1.2 x ULN | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2
  Monocytes/Leukocytes >1.2 x ULN: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 2 | 2 | 5 | 1 | 11
  Monocytes/Leukocytes >1.2 x ULN | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 1 | 1 | 1
  Bilirubin >1.5 x ULN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Direct Bilirubin >1.5 x ULN: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 3 | 5 | 1 | 11
  Direct Bilirubin >1.5 x ULN | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
  Aspartate Aminotransferase >3.0 x ULN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea >1.3 x ULN | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urate >1.2 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Creatine Kinase >2.0 x ULN: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatine Kinase >2.0 x ULN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C Reactive Protein >1.1 x ULN: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 3 | 3 | 6 | 6 | 6 | 3 | 11
  C Reactive Protein >1.1 x ULN | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 2 | 3 | 2 | 0
  Bicarbonate >1.1 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  D-Dimer >1.5 x ULN | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 1 | 1 | 2 | 0 | 1
  Fibrinogen >1.25 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Specific Gravity <1.003: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 3 | 5 | 1 | 11
  Specific Gravity <1.003 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Specific Gravity >1.030: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 3 | 5 | 1 | 11
  Specific Gravity >1.030 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  pH >8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Ketones ≥1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 0 | 0 | 1
  URINE Protein ≥1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  URINE Hemoglobin ≥1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 5 | 5 | 6 | 3 | 16
  URINE Hemoglobin ≥1 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1
  Urobilinogen ≥1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1
  URINE Bilirubin ≥1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Nitrite ≥1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Leukocyte Esterase ≥1: number analyzed (Participants) | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 4 | 4 | 1 | 2 | 8
  Leukocyte Esterase ≥1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Vital Signs Meeting Categorical Criteria
Description: Supine blood pressure and pulse rate were measured. Categorical classes for vital signs of potential clinical concerns were defined as followed: systolic blood pressure (SBP) <90 millimeters of mercury (mmHg); diastolic blood pressure (DBP) <50 mmHg; pulse rate <40 beats per minute (bpm); pulse rate >120 bpm, and increase from baseline in SBP ≥30 mmHg; decrease from baseline in SBP ≥30 mmHg; increase from baseline in DBP ≥20 mmHg; decrease from baseline in DBP ≥20 mmHg. Baseline was defined as the mean of the replicated predose (0 hour) measurement on Day 1.
Time Frame: as for outcome 2
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16
Participants
  Pulse rate <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 3 | 0
  Pulse rate >120 bpm | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP <50 mmHg | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  DBP: increase from baseline ≥20 mmHg | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 1 | 0
  DBP: decrease from baseline ≥20 mmHg | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP <90 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP: increase from baseline ≥30 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP: decrease from baseline ≥30 mmHg | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Electrocardiograms (ECGs) Meeting Categorical Criteria
Description: Number of participants with ECG findings meeting the following criteria: time between the onset of atrial depolarization and onset of ventricular depolarization (PR interval) ≥300 msec; time from ECG Q-wave to the end of the S wave corresponding to ventricular depolarization (QRS duration) ≥140 msec; correct time from ECG Q-wave to the end of the T wave corresponding to electrical systole for heart rate using Fridericia's formula (QTcF interval): ≥450 to <480 msec; QTcF interval ≥480 to <500 msec; QTcF interval: ≥500 msec; PR interval percent change from baseline (≥25/50%): ≥25% if baseline >200 msec or ≥ 50% if baseline ≤200 msec; QRS duration percent change from baseline ≥50%; QTcF interval change from baseline: >30 to ≤60 msec; QTcF interval change from baseline >60 msec. Baseline was defined as the average of the triplicate predose recordings collected at 0 hour on Day 1.
Time Frame: Baseline (Study Day 1, predose), Study Days 1 (postdose), 2, 4, 6, 8, 11, 22, 36 (end of study visit for IV treatment cohorts) and 71 (end of study visit for SC treatment cohorts).
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16
Participants
  PR interval ≥300 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR interval: percent change from baseline ≥25/50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS duration ≥140 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS duration: percent change from baseline ≥50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval: ≥450 to <480 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval: ≥480 to <500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval ≥500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval change from baseline: >30 msec to ≤60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval change from baseline: >60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-06755347 Following Single IV Dose
Description: Cmax was the highest concentration observed directly from data
Time Frame: Hours 0, 1, 3, 5, 8, 12, 24, 48, 72, 120, and 168 for every cohort, hour 36 for Cohorts 1 and 2, Days 15, 22, 29, and 36 for Cohorts 3-6, hours 3.5, 4, and 6 for Cohorts 5 and 6.
Population: All randomized participants who received at least 1 dose of PF-06755347 and had at least 1 of the PK parameters of interest. No results were reported for 16 participants who received placebo because participants didn't receive the investigational product and had no PK parameter of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (ug/mL)
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
micrograms/milliliter (ug/mL) | 0.1123 (18) | 0.4462 (20) | 1.654 (10) | 4.700 (9) | 24.72 (21) | 12.36 (9)

6. Secondary Outcome: Cmax of PF-06755347 Following Single SC Dose
Description: Cmax was the highest concentration observed directly from data
Time Frame: Hours 0, 12, 24, 48, 72, 120, and 168, and Days 5, 11, 15, 22, 29, 36, 50 and 71.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 3
ug/mL | 0.8946 (25) | 1.374 (68) | 2.641 (40) | 5.678 (15) | 5.276 (47)

7. Secondary Outcome: Dose Normalized Cmax (Cmax(dn)) of PF-06755347 Following Single IV Dose
Description: Cmax(dn) = Cmax/Dose
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL/(miligrams/kilogram [mg/kg])
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
ug/mL/(miligrams/kilogram [mg/kg]) | 11.23 (18) | 14.88 (20) | 16.54 (10) | 15.69 (9) | 24.72 (21) | 17.68 (9)

8. Secondary Outcome: Cmax(dn) of PF-06755347 Following Single SC Dose
Description: Cmax(dn) = Cmax/Dose
Time Frame: Hours 0, 12, 24, 48, 72, 120, and 168, and Days 5, 11, 15, 22, 29, 36, 50 and 71.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL/(mg/kg)
Arm/Group | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 3
ug/mL/(mg/kg) | 0.03579 (25) | 0.02748 (68) | 0.02641 (40) | 0.02842 (15) | 5.276 (0.01758)

9. Secondary Outcome: Time for Cmax (Tmax) of PF-06755347 Following Single IV Dose
Description: Tmax was the time to reach maximum observed plasma concentration, which was observed directly from data as time of first occurrence.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
hours | 1.270 [1.22 to 1.30] | 1.050 [1.05 to 1.08] | 1.180 [1.17 to 1.18] | 1.180 [1.18 to 1.18] | 1.170 [1.17 to 3.30] | 3.020 [1.00 to 3.03]

10. Secondary Outcome: Tmax of PF-06755347 Following Single SC Dose
Description: as for outcome 9
Time Frame: Hours 0, 12, 24, 48, 72, 120, and 168, and Days 5, 11, 15, 22, 29, 36, 50 and 71.
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 3
hours | 48.00 [48.00 to 72.00] | 48.00 [48.00 to 48.90] | 60.05 [48.00 to 96.00] | 48.00 [24.00 to 96.00] | 72.00 [48.00 to 120.00]

11. Secondary Outcome: Area Under the Concentration-time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-06755347 Following Single IV Dose
Description: AUClast was determined using linear/Log trapezoidal method
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter (ug*hr/mL)
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
micrograms*hour/milliliter (ug*hr/mL) | 1.395 (70) | 10.51 (30) | 45.18 (9) | 156.4 (7) | 511.8 (29) | 316.2 (3)

12. Secondary Outcome: AUClast of PF-06755347 Following Single SC Dose
Description: AUClast was determined using linear/Log trapezoidal method
Time Frame: Hours 0, 12, 24, 48, 72, 120, and 168, and Days 5, 11, 15, 22, 29, 36, 50 and 71.
Population: All randomized participants who received at least one dose of PF-06755347 and had at least 1 of the PK parameters of interest. No results were reported for 16 participants who received placebo because participants didn't receive the investigational product and had no PK parameter of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 3
ug*hr/mL | 125.4 (12) | 230.2 (42) | 428.7 (24) | 859.5 (13) | 977.6 (30)

13. Secondary Outcome: Dose Normalized AUClast (AUClast(dn)) of PF-06755347 Following Single IV Dose
Description: AUClast(dn) = AUClast/Dose
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL/(mg/kg)
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
ug*hr/mL/(mg/kg) | 139.5 (70) | 349.8 (30) | 451.8 (9) | 521.1 (7) | 511.8 (29) | 451.8 (3)

14. Secondary Outcome: AUClast(dn) of PF-06755347 Following Single SC Dose
Description: AUClast(dn) = AUClast/Dose
Time Frame: Hours 0, 12, 24, 48, 72, 120, and 168, and Days 5, 11, 15, 22, 29, 36, 50 and 71.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL/(mg/kg)
Arm/Group | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 3
ug*hr/mL/(mg/kg) | 5.010 (13) | 4.603 (42) | 4.287 (24) | 4.297 (13) | 3.263 (30)

15. Secondary Outcome: Area Under the Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of PF-06755347 Following Single IV Dose
Description: AUClast + (Clast*/kel), where Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis and kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 5
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 3 | 2
ug*hr/mL |  | 12.52 (25) | 49.35 (10) | 162.7 (8) | 569.7 (29) | NA (NA) — Geo mean was not calculated due to <3 contributes.

16. Secondary Outcome: AUCinf of PF-06755347 Following Single SC Dose
Description: as for outcome 15
Time Frame: Hours 0, 12, 24, 48, 72, 120, and 168, and Days 5, 11, 15, 22, 29, 36, 50 and 71.
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC
Number analyzed (Participants) | 3 | 5 | 6 | 5 | 3
ug*hr/mL | 133.2 (10) | 234.7 (42) | 440.1 (25) | 861.3 (15) | 988.8 (30)

17. Secondary Outcome: Dose Normalized AUCinf (AUCinf(dn)) of PF-06755347 Following Single IV Dose
Description: AUCinf(dn) = AUCinf/Dose
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL/mg
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 3 | 2
ug*hr/mL/mg |  | 417.5 (25) | 493.5 (10) | 541.9 (8) | 569.7 (29) | NA (NA) — Geo mean was not calculated due to <3 contributes.

18. Secondary Outcome: AUCinf(dn) of PF-06755347 Following Single SC Dose
Description: AUCinf(dn) = AUCinf/Dose
Time Frame: Hours 0, 12, 24, 48, 72, 120, and 168, and Days 5, 11, 15, 22, 29, 36, 50 and 71.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL/mg
Arm/Group | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC
Number analyzed (Participants) | 3 | 5 | 6 | 5 | 3
ug*hr/mL/mg | 5.323 (11) | 4.695 (42) | 4.401 (25) | 4.305 (15) | 3.295 (30)

19. Secondary Outcome: Terminal Half-life (t½) of PF-06755347 Following Single IV Dose
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. t½ = Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 5
Population: All randomized participants who received at least one dose and had at least 1 of the PK parameters of interest. All randomized participants who received at least one dose and had at least 1 of the PK parameters of interest. No results were reported for 16 participants who received placebo because participants didn't receive the investigational product and had no PK parameter of interest.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 3 | 2
hours |  | 34.20 (7.3082) | 51.10 (4.7624) | 77.17 (0.40415) | 70.90 (12.150) | NA (NA) — Geo mean was not calculated due to <3 contributes.

20. Secondary Outcome: t½ of PF-06755347 Following Single SC Dose
Description: as for outcome 19
Time Frame: Hours 0, 12, 24, 48, 72, 120, and 168, and Days 5, 11, 15, 22, 29, 36, 50 and 71.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC
Number analyzed (Participants) | 3 | 5 | 6 | 5 | 3
hours | 94.13 (32.843) | 135.6 (56.409) | 82.88 (19.498) | 100.1 (18.940) | 139.3 (9.8658)

21. Secondary Outcome: Clearance (CL) of PF-06755347 Following Single IV Dose
Description: CL = Dose/AUCinf Steady state total body clearance equals infusion rate (zero order) divided by steady state plasma concentration of study drug.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr/kg
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 3 | 2
L/hr/kg |  | 0.002397 (25) | 0.002027 (10) | 0.001846 (8) | 0.001758 (29) | NA (NA) — Geo mean was not calculated due to <3 contributes.

22. Secondary Outcome: Apparent Clearance (CL/F) of PF-06755347 Following Single SC Dose
Description: CL/F = Dose/AUCinf Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Hours 0, 12, 24, 48, 72, 120, and 168, and Days 5, 11, 15, 22, 29, 36, 50 and 71.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC
Number analyzed (Participants) | 3 | 5 | 6 | 5 | 3
L/hr | 0.1876 (11) | 0.2128 (42) | 0.2272 (25) | 0.2321 (15) | 0.3036 (30)

23. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody to PF-06755347
Description: Human serum samples were analyzed for the presence or absence of anti-PF-06755347 antibodies (ADA) following a tiered approach of screening, confirmation and titer determination, using an electrochemiluminescent (ECL) immunoassay. Baseline was the measurement on Day -1.
Time Frame: Baseline, Study Days 8, 15, and 36 for all treatment cohorts plus Day 71 for SC treatment cohorts
Population: All participants who received at least 1 dose of study medication. Number of participants analyzed represents the total number of participants in each treatment group in the analysis population for this outcome measure. Number analyzed represents the number of participants who had reportable results for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16
Participants
  Baseline postive ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3
  Day 8 positive ADA: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 3 | 16
  Day 8 positive ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Day 15 positive ADA: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1 | 2 | 2 | 6 | 5 | 4 | 3 | 15
  Day 15 positive ADA | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Day 36 positive ADA: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 2 | 2 | 6 | 5 | 5 | 3 | 15
  Day 36 positive ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Day 71 positive ADA: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 6 | 5 | 3 | 8
  Day 71 positive ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1

24. Secondary Outcome: Change From Baseline in Interferon Gamma (IFN-γ ) at Scheduled Timepoints
Description: IFN-γ was one of the 3 cytokine biomarkers explored in the study. Baseline was defined as the average of measurement on Day -1 and pre-dose (0 hours) measurement on Day 1.
Time Frame: Day -1, hours 0, 5, 12, 24, 48, 72 for all treatment cohorts. Hours 1 (or end of infusion), 8, and 120 and Days 11 and 29 for IV treatment cohorts; Days 5, 8, 15, 36 and 71 for SC treatment cohorts.
Population: All enrolled participants treated who had at least 1 measurement of the exploratory endpoints of interest. Number of participants analyzed represents the total number of participants in each treatment group in the analysis population for this outcome measure. Number analyzed represents the number of participants who had reportable results for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanograms per liter (ng/L)
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16
nanograms per liter (ng/L)
  Day 1: 1 hour post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 1 | 0 | 0 | 10
  Day 1: 1 hour post-dose | -0.303 (0.0950) | -3.230 (5.0126) | -0.337 (0.5686) | 3.903 (3.7969) | 20.240 (14.2259) | 26.157 (17.0904) | -0.423 (0.2454) | -0.145 (0.8771) | -0.030 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | -0.554 (0.4981)
  Day 1: 3 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 1 | 0 | 0 | 10
  Day 1: 3 hours post-dose | -0.440 (0.7134) | -0.293 (3.4514) | 24.490 (22.6078) | 50.667 (29.7923) | 292.287 (233.1423) | 250.257 (301.3490) | -0.403 (0.4239) | 0.295 (0.8520) | 0.330 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | -0.448 (0.4631)
  Day 1: 5 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 6 | 6 | 3 | 16
  Day 1: 5 hours post-dose | 0.383 (1.2687) | -1.227 (5.1897) | 16.790 (13.5079) | 21.467 (11.4311) | 160.287 (157.2547) | 41.575 (15.6624) | 0.223 (1.2471) | 4.155 (10.1704) | 4.403 (5.7437) | 53.540 (65.4359) | 14.793 (7.5312) | -0.337 (0.7686)
  Day 1: 8 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 1 | 0 | 0 | 5
  Day 1: 8 hours post-dose |  |  |  |  | 86.700 (NA) — Standard deviaiton is not calculable for 1 value. | 9.975 (1.5910) | 1.373 (1.9731) | 5.012 (12.0362) | 14.400 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | -0.422 (0.4181)
  Day 1: 12 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 6 | 6 | 3 | 11
  Day 1: 12 hours post-dose |  |  |  |  | 32.100 (NA) — Standard deviaiton is not calculable for 1 value. | 4.125 (7.9550) | 2.477 (2.8330) | 4.230 (7.9003) | 11.207 (5.8049) | 12.345 (4.5839) | 8.327 (6.7983) | -0.155 (0.8139)
  Day 2: 24 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 6 | 6 | 3 | 16
  Day 2: 24 hours post-dose | 0.430 (2.1622) | -1.750 (4.2354) | -0.403 (0.8138) | -0.317 (0.3868) | -12.533 (21.7084) | 21.075 (44.2295) | 2.340 (3.1990) | 2.402 (2.8296) | 3.322 (2.1890) | 3.283 (1.6786) | -3.257 (9.1184) | 1.027 (3.3372)
  Day 3: 48 hours post-dose | 5.400 (11.9840) | -4.707 (8.0587) | -0.083 (0.1893) | -0.497 (0.4405) | -8.733 (15.1266) | 2.663 (14.6931) | 2.820 (5.9672) | 1.333 (4.4335) | 2.937 (3.8441) | 1.563 (0.9806) | -5.300 (9.5979) | 12.843 (50.7623)
  Day 4: 72 hours post-dose | 2.877 (8.4727) | -4.893 (8.0609) | -0.433 (1.0587) | -0.363 (0.3702) | -15.327 (26.5466) | -3.660 (5.9789) | 1.197 (2.2445) | -2.492 (8.4374) | 0.968 (2.5824) | 0.552 (1.0780) | -6.063 (10.1365) | 27.946 (111.802)
  Day 5: 96 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 3 | 6
  Day 5: 96 hours post-dose |  |  |  |  |  |  |  |  | 0.558 (2.0766) | 8.516 (15.1062) | -6.123 (10.0962) | 1.118 (1.5380)
  Day 8: 168 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 3 | 16
  Day 8: 168 hours post-dose | -0.817 (2.8587) | -8.260 (13.1193) | -0.487 (0.7658) | -0.230 (0.3279) | -16.247 (28.1401) | -3.290 (3.3698) | -0.160 (1.5159) | -3.900 (12.0196) | -2.040 (3.6754) | -0.344 (0.9542) | -5.457 (9.9449) | 1.006 (3.8100)
  Day 15: 336 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1 | 2 | 2 | 6 | 5 | 4 | 3 | 15
  Day 15: 336 hours post-dose | -0.413 (3.6272) | -10.640 (16.1897) | 1.240 (1.0792) | -0.050 (0.5766) | 0.000 (NA) — Standard deviaiton is not calculable for 1 value. | 0.900 (9.2772) | 0.005 (0.2475) | -5.550 (12.2071) | -1.864 (3.5365) | -0.133 (0.9903) | -2.833 (4.3584) | 0.713 (5.8229)
  Day 36: 840 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 2 | 2 | 6 | 5 | 5 | 3 | 14
  Day 36: 840 hours post-dose | 25.507 (44.6205) | -11.603 (18.4042) | 0.510 (0.7119) | 0.097 (0.3807) |  | -0.960 (7.2832) | 2.985 (2.8214) | -5.598 (11.5371) | 5.650 (12.4743) | -0.188 (1.5621) | -4.397 (7.4304) | 1.276 (3.1066)
  Day 71: 1680 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 6 | 5 | 3 | 8
  Day 71: 1680 hours post-dose |  |  |  |  |  |  | 0.853 (0.2040) | -5.755 (12.4057) | -2.120 (4.0010) | 0.082 (1.6527) | -4.830 (10.8140) | 1.019 (0.8362)

25. Secondary Outcome: Change From Baseline in Tumor Necrosis Factor Alpha (TNFα) at Scheduled Timepoints
Description: TNFα was one of the 3 cytokine biomarkers explored in the study. Baseline was defined as the average of measurement on Day -1 and pre-dose (0 hours) measurement on Day 1.
Time Frame: as for outcome 24
Population: All enrolled subjects treated who had at least 1 measurement of the exploratory endpoints of interest. "Number Analyzed" in each row will be 0 if no participant had at least 1 measurement of the exploratory endpoints of interest within the specified timeframe.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16
ng/L
  Day 1: 1 hour post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 1 | 0 | 0 | 10
  Day 1: 1 hour post-dose | -0.0500 (0.06000) | -0.0667 (0.31565) | 0.6533 (0.83032) | 4.8733 (3.27147) | 59.7100 (34.37035) | 38.5200 (29.69790) | -0.0250 (0.06051) | 0.0048 (0.06199) | 0.1200 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | 0.0055 (0.11117)
  Day 1: 3 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 1 | 0 | 0 | 10
  Day 1: 3 hours post-dose | -0.1100 (0.21932) | 0.4567 (0.21939) | 10.7767 (10.67258) | 20.4567 (7.74517) | 217.9767 (78.32721) | 97.4267 (89.31240) | 0.0327 (0.08016) | 0.1905 (0.27975) | 0.3600 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | 0.0198 (0.12203)
  Day 1: 5 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 6 | 6 | 3 | 16
  Day 1: 5 hours post-dose | -0.0833 (0.08505) | 0.1333 (0.27062) | 5.8100 (3.05779) | 9.0900 (1.62613) | 49.6433 (18.57913) | 15.6900 (4.25678) | 0.0673 (0.10808) | 0.5760 (1.36848) | 0.3422 (0.43494) | 10.4592 (16.00977) | 1.7770 (0.92867) | -0.1024 (0.08281)
  Day 1: 8 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 1 | 0 | 0 | 5
  Day 1: 8 hours post-dose |  |  |  |  | 23.8900 (NA) — Standard deviaiton is not calculable for 1 value. | 5.6750 (2.41123) | 0.3103 (0.37419) | 0.6442 (1.36307) | 1.7800 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | -0.1326 (0.13676)
  Day 1: 12 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 6 | 6 | 3 | 11
  Day 1: 12 hours post-dose |  |  |  |  | 11.0900 (NA) — Standard deviaiton is not calculable for 1 value. | 2.7700 (1.41421) | 0.4367 (0.48959) | 0.4453 (0.65376) | 1.1792 (0.71557) | 1.7025 (0.71450) | 1.3270 (0.18793) | -0.1489 (0.13550)
  Day 2: 24 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 6 | 6 | 3 | 16
  Day 2: 24 hours post-dose | 0.2567 (0.06110) | 0.0567 (0.31501) | 1.3067 (0.25325) | 0.8700 (0.09644) | 2.8000 (1.25790) | 1.6150 (1.77484) | 0.1383 (0.05777) | 0.3792 (0.53143) | 0.9425 (0.50586) | 1.0875 (0.40787) | 0.7370 (0.19120) | 0.0585 (0.13732)
  Day 3: 48 hours post-dose | 0.2200 (0.30447) | 0.0333 (0.21362) | 0.5967 (0.17559) | 0.0933 (0.54151) | 0.4967 (0.30022) | 0.7533 (1.52998) | 0.0883 (0.06213) | 0.1830 (0.20827) | 0.5225 (0.24791) | 0.5575 (0.24078) | 0.4237 (0.06199) | 0.0784 (0.29068)
  Day 4: 72 hours post-dose | 0.0433 (0.44004) | -0.0167 (0.39954) | 0.2767 (0.32929) | -0.1467 (0.32470) | 0.0900 (0.22539) | 0.7100 (1.04159) | 0.0227 (0.12889) | 0.1182 (0.20360) | 0.2665 (0.14113) | 0.1608 (0.17623) | 0.3293 (0.11039) | 0.2039 (0.73037)
  Day 5: 96 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 3 | 6
  Day 5: 96 hours post-dose |  |  |  |  |  |  |  |  | 0.1820 (0.10060) | 0.1644 (0.14800) | 0.2643 (0.06914) | -0.0080 (0.10568)
  Day 8: 168 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 3 | 16
  Day 8: 168 hours post-dose | -0.1600 (0.38974) | -0.3633 (0.52205) | 0.1867 (0.54647) | -0.0667 (0.43730) | 0.0267 (0.31342) | 0.2233 (0.32130) | -0.0350 (0.12758) | 0.0383 (0.17292) | -0.0317 (0.17725) | 0.0098 (0.04696) | 0.1697 (0.05604) | 0.0237 (0.20192)
  Day 15: 336 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1 | 2 | 2 | 6 | 5 | 4 | 3 | 15
  Day 15: 336 hours post-dose | -0.1833 (0.37873) | -0.4133 (0.56722) | 0.5033 (0.71501) | -0.1233 (0.10017) | 0.2300 (NA) — Standard deviaiton is not calculable for 1 value. | -0.5810 (0.96308) | 0.1685 (0.26092) | 0.2715 (0.36900) | 0.0280 (0.16664) | 0.0310 (0.12138) | 0.1297 (0.30426) | 0.0909 (0.49582)
  Day 36: 840 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 2 | 2 | 6 | 5 | 5 | 3 | 14
  Day 36: 840 hours post-dose | 0.3233 (0.21733) | -0.5767 (0.99470) | 0.4867 (0.96500) | 0.2633 (0.63129) |  | -1.2265 (0.15910) | 0.0650 (0.41154) | 0.4748 (0.44527) | 0.2776 (0.56067) | -0.1340 (0.19649) | -0.0040 (0.02330) | -0.0090 (0.85788)
  Day 71: 840 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 6 | 5 | 3 | 8
  Day 71: 840 hours post-dose |  |  |  |  |  |  | 0.1363 (0.25455) | 0.5913 (0.28774) | -0.0340 (0.25211) | -0.1698 (0.20600) | 0.1327 (0.19433) | -0.0820 (0.24109)

26. Secondary Outcome: Change From Baseline in Interleukin 6 (IL-6) at Scheduled Timepoints
Description: IL-6 was one of the 3 cytokine biomarkers explored in the study. Baseline was defined as the average of measurement on Day -1 and pre-dose (0 hours) measurement on Day 1.
Time Frame: as for outcome 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16
ng/L
  Day 1: 1 hour post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 1 | 0 | 0 | 10
  Day 1: 1 hour post-dose | 0.0177 (0.03060) | -0.0207 (0.08003) | 0.0743 (0.12009) | 0.9653 (1.35472) | 0.6757 (0.80530) | 2.1110 (2.86966) | 0.0000 (0.00000) | 0.2665 (0.38316) | 0.1410 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | 0.0120 (0.07478)
  Day 1: 3 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 1 | 0 | 0 | 10
  Day 1: 3 hours post-dose | 0.7137 (0.53129) | 0.3280 (0.33207) | 4.7613 (5.00708) | 24.9907 (28.82106) | 1261.782 (1377.243) | 365.8777 (534.9345) | 0.2863 (0.13785) | 2.3943 (2.26382) | 1.1740 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | 0.3684 (0.77453)
  Day 1: 5 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 6 | 6 | 3 | 16
  Day 1: 5 hours post-dose | 0.8893 (0.97631) | 0.6083 (0.46302) | 5.4180 (6.21463) | 10.7307 (5.75904) | 817.4487 (952.5663) | 16.1545 (9.43210) | 0.2970 (0.31973) | 2.8793 (2.33024) | 1.7130 (2.18458) | 53.7213 (107.2734) | 11.1390 (16.70153) | 0.2653 (0.48087)
  Day 1: 8 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 1 | 0 | 0 | 5
  Day 1: 8 hours post-dose |  |  |  |  | 35.2980 (NA) — Standard deviaiton is not calculable for 1 value. | 0.3100 (0.65620) | 0.4090 (0.31213) | 3.1483 (4.27777) | 1.7440 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | 0.6368 (0.62657)
  Day 1: 12 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 6 | 6 | 3 | 11
  Day 1: 12 hours post-dose |  |  |  |  | 6.4480 (NA) — Standard deviaiton is not calculable for 1 value. | 0.1375 (0.81529) | 0.7460 (0.42248) | 3.3927 (1.80711) | 1.9242 (2.23190) | 1.2097 (0.72824) | 0.6550 (0.33707) | 0.3799 (0.63486)
  Day 2: 24 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 6 | 6 | 3 | 16
  Day 2: 24 hours post-dose | 0.0817 (0.14145) | 0.1917 (0.24744) | 0.2260 (0.23010) | 0.1040 (0.09938) | 0.8647 (0.93571) | -0.0495 (0.55084) | 0.4147 (0.71822) | 3.5448 (3.52636) | 0.2730 (0.29167) | 0.0957 (0.13221) | 1.3477 (2.13897) | 0.1433 (0.20404)
  Day 3: 48 hours post-dose | 0.3813 (0.66049) | -0.0063 (0.04087) | 0.0927 (0.10203) | 0.0120 (0.4405) | -0.0667 (0.11547) | -0.0937 (0.30933) | 0.5713 (0.98958) | 0.2855 (0.60079) | 2.1285 (4.43835) | 0.0155 (0.03797) | 0.5043 (0.80624) | 0.0974 (0.35056)
  Day 4: 72 hours post-dose | 0.3947 (0.68358) | 0.3010 (0.30959) | -0.0087 (0.01250) | 0.0960 (0.16628) | 0.6127 (1.06117) | -0.1297 (0.26905) | 0.1830 (0.16928) | 0.1143 (0.22064) | 0.2382 (0.53605) | 0.1062 (0.13652) | -0.0157 (0.02714) | 0.1368 (0.81459)
  Day 5: 96 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 3 | 6
  Day 5: 96 hours post-dose |  |  |  |  |  |  |  |  | 0.0834 (0.73122) | 1.7690 (3.78958) | -0.0277 (0.04792) | 0.0000 (0.0000)
  Day 8: 168 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 3 | 16
  Day 8: 168 hours post-dose | 0.0787 (0.13625) | -0.0310 (0.05369) | 0.0727 (0.06972) | 0.0000 (0.0000) | 0.0070 (0.23658) | -0.1203 (0.27872) | 0.0000 (0.00000) | 0.0780 (0.10187) | 0.0100 (0.81680) | 0.0284 (0.06350) | 0.0180 (0.03118) | -0.0282 (0.56396)
  Day 15: 336 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1 | 2 | 2 | 6 | 5 | 4 | 3 | 15
  Day 15: 336 hours post-dose | 0.0847 (0.11301) | 0.1570 (0.27193) | 0.1563 (0.15264) | 2.1150 (3.50770) | 0.0000 (NA) — Standard deviaiton is not calculable for 1 value. | 0.5620 (0.79479) | 0.0000 (0.0000) | 0.0298 (0.08751) | -0.0998 (0.40069) | 0.0000 (0.0000) | 0.2797 (0.48440) | -0.0737 (0.43828)
  Day 36: 840 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 2 | 2 | 6 | 5 | 5 | 3 | 14
  Day 36: 840 hours post-dose | 0.7927 (1.36082) | -0.0247 (0.04272) | 0.3590 (0.27029) | 0.0340 (0.05889) |  | 0.0000 (0.0000) | 0.0105 (0.01485) | -0.0047 (0.01143) | 0.1396 (0.23005) | 0.0774 (0.17307) | 0.0710 (0.12298) | 0.0861 (0.15271)
  Day 71: 1680 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 6 | 5 | 3 | 8
  Day 71: 1680 hours post-dose |  |  |  |  |  |  | 0.0000 (0.0000) | 0.0255 (0.07700) | -0.0758 (0.61407) | 0.0000 (0.0000) | 0.2030 (0.35161) | 0.0539 (0.16145)

27. Secondary Outcome: Change From Baseline in Complement 3a (C3a) at Scheduled Timepoints
Description: C3a was one of the 3 complement components/biomarkers explored in the study. Baseline was defined as the average of measurement on Day -1 and pre-dose (0 hours) measurement on Day 1.
Time Frame: as for outcome 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: micrograms per liter (mcg/L)
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16
micrograms per liter (mcg/L)
  Day 1: 1 hour post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 1 | 0 | 0 | 10
  Day 1: 1 hour post-dose | 2234.0 (2663.07) | 0.0 (0.00) | 1570.0 (795.05) | 730.0 (1889.87) | 2680.7 (2327.03) | 4310.0 (3997.14) | 260.0 (450.33) | 131.8 (317.57) | 0.0 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | -425.1 (779.62)
  Day 1: 3 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 1 | 0 | 0 | 10
  Day 1: 3 hours post-dose | 0.0 (0.00) | 0.0 (0.00) | -133.3 (675.45) | -827.0 (1293.35) | 1017.0 (1761.50) | 360.0 (2941.56) | -13.3 (23.09) | 1138.7 (2152.68) | 0.0 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | -364.0 (937.82)
  Day 1: 5 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 6 | 6 | 3 | 16
  Day 1: 5 hours post-dose | 0.0 (0.00) | 0.0 (0.00) | 1219.7 (2513.81) | -1214.0 (1129.48) | 33.7 (58.31) | -115.5 (3741.30) | 13.3 (23.09) | 188.5 (296.99) | 1348.5 (1359.62) | -170.2 (796.82) | 1093.7 (1681.60) | -162.0 (767.87)
  Day 1: 8 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 1 | 0 | 0 | 5
  Day 1: 8 hours post-dose |  |  |  |  | 0.0 (NA) — Standard deviaiton is not calculable for 1 value. | -430.5 (3295.82) | -70.0 (121.24) | 541.8 (844.36) | 0.0 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | -176.0 (393.55)
  Day 1: 12 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 6 | 6 | 3 | 11
  Day 1: 12 hours post-dose |  |  |  |  | 0.0 (NA) — Standard deviaiton is not calculable for 1 value. | 1650.0 (3691.10) | -173.7 (300.80) | 705.2 (1132.91) | 518.3 (752.66) | -583.5 (1326.10) | 440.0 (762.10) | 569.3 (1040.58)
  Day 2: 24 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 6 | 6 | 3 | 16
  Day 2: 24 hours post-dose | 0.0 (0.00) | 33.7 (58.31) | 3626.3 (4819.80) | -1394.0 (1422.73) | 507.0 (878.15) | -1425.5 (1888.68) | 526.7 (1388.08) | 588.5 (1225.78) | 383.3 (890.52) | -548.5 (1846.32) | -76.7 (132.79) | -187.4 (1055.28)
  Day 3: 48 hours post-dose | 0.0 (0.00) | 10.3 (17.90) | 516.7 (1030.55) | -937.3 (2577.06) | 737.0 (1276.52) | -333.7 (1803.48) | -173.7 (300.80) | 210.2 (711.62) | 1418.5 (2194.12) | -640.5 (1839.01) | 330.0 (571.58) | 174.3 (1669.50)
  Day 4: 72 hours post-dose | 83.7 (144.9) | 80.3 (139.14) | -170.0 (810.19) | -1561.0 (1700.71) | 0.0 (0.00) | -757.0 (1336.62) | -53.3 (92.38) | 65.0 (581.79) | 295.2 (739.73) | -1133.7 (1614.09) | 710.0 (1229.76) | -77.6 (766.58)
  Day 5: 96 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 3 | 6
  Day 5: 96 hours post-dose |  |  |  |  |  |  |  |  | 475.8 (777.97) | -252.2 (2190.36) | -346.7 (600.44) | 788.2 (2632.47)
  Day 8: 168 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 3 | 16
  Day 8: 168 hours post-dose | 407.0 (704.94) | 0.0 (0.00) | -240.7 (1064.66) | -1120.7 (2039.85) | 403.7 (699.17) | -407.0 (2048.41) | -173.7 (300.80) | 530.2 (822.22) | 876.7 (993.91) | -1078.2 (1941.86) | 383.3 (663.95) | 262.4 (1096.43)
  Day 15: 336 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1 | 2 | 2 | 6 | 5 | 4 | 3 | 15
  Day 15: 336 hours post-dose | 0.0 (0.00) | 0.0 (0.00) | 519.7 (2234.46) | -780.3 (594.56) | 0.0 (NA) — Standard deviaiton is not calculable for 1 value. | 129.5 (1075.51) | -260.5 (368.40) | 1410.5 (2078.58) | -536.4 (602.28) | -688.0 (2313.92) | 693.3 (1200.89) | -70.7 (1343.24)
  Day 36: 840 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 2 | 2 | 6 | 5 | 5 | 3 | 14
  Day 36: 840 hours post-dose | 1727.3 (1545.92) | 0.0 (0.00) | 1960.0 (2817.68) | -1561.0 (1700.71) |  | -656.0 (35.36) | -260.5 (368.40) | 567.2 (729.62) | 1062.2 (2324.85) | -1298.4 (1672.16) | 693.3 (1200.89) | 470.0 (3018.14)
  Day 71: 1680 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 6 | 5 | 3 | 8
  Day 71: 1680 hours post-dose |  |  |  |  |  |  | 1713.3 (3428.69) | 1830.8 (1654.01) | 2330.3 (3100.19) | -1734.6 (1602.72) | 156.7 (271.35) | 436.1 (1343.41)

28. Secondary Outcome: Change From Baseline in Complement 5a (C5a) at Scheduled Timepoints
Description: C5a was one of the 3 complement components/biomarkers explored in the study. Baseline was defined as the average of measurement on Day -1 and pre-dose (0 hours) measurement on Day 1.
Time Frame: as for outcome 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16
mcg/L
  Day 1: 1 hour post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 1 | 0 | 0 | 10
  Day 1: 1 hour post-dose | 0.623 (0.4709) | -0.167 (1.6862) | 0.213 (0.2676) | -0.283 (0.6417) | -0.627 (0.2098) | -0.613 (0.0643) | 0.083 (0.1193) | -0.283 (0.6940) | 5.300 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | -0.183 (0.8073)
  Day 1: 3 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 1 | 0 | 0 | 10
  Day 1: 3 hours post-dose | 0.870 (0.2343) | -0.057 (0.9869) | -0.040 (0.2862) | -0.983 (0.7184) | -0.827 (0.4311) | -0.655 (0.0071) | 0.023 (0.0681) | -0.153 (0.4864) | 11.300 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | -0.219 (1.3316)
  Day 1: 5 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 6 | 6 | 3 | 16
  Day 1: 5 hours post-dose | -0.027 (0.0379) | 4.413 (9.3654) | -0.067 (0.3150) | -1.140 (1.2813) | -0.317 (0.3281) | -0.485 (0.2475) | 0.127 (0.1115) | -0.183 (0.4491) | 4.102 (6.1943) | -0.177 (0.7212) | 0.410 (0.3996) | -0.176 (1.0820)
  Day 1: 8 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 1 | 0 | 0 | 5
  Day 1: 8 hours post-dose |  |  |  |  | 0.710 (NA) — Standard deviaiton is not calculable for 1 value. | -0.445 (0.3041) | 0.013 (0.0231) | -0.275 (0.7237) | 7.700 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | -0.130 (0.4181)
  Day 1: 12 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 6 | 6 | 3 | 11
  Day 1: 12 hours post-dose |  |  |  |  | -0.680 (NA) — Standard deviaiton is not calculable for 1 value. | -0.605 (0.0778) | 0.210 (0.3637) | -0.220 (0.7804) | -4.413 (6.3713) | 0.035 (0.7219) | 0.043 (0.4466) | -0.044 (0.6347)
  Day 2: 24 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 6 | 6 | 3 | 16
  Day 2: 24 hours post-dose | 0.907 (0.6881) | 0.730 (2.6751) | 0.003 (0.6153) | 2.713 (4.5502) | 3.717 (3.8882) | -0.670 (0.0141) | 0.190 (0.3291) | -0.233 (0.7781) | 0.767 (9.8244) | 0.425 (0.8435) | -0.380 (0.5027) | -0.015 (0.5437)
  Day 3: 48 hours post-dose | 0.987 (0.9901) | 1.077 (3.6656) | 0.360 (0.4004) | 0.833 (3.0087) | 2.043 (2.4110) | -0.403 (0.3194) | 0.197 (0.3406) | -0.062 (0.8170) | -0.142 (8.3021) | -0.235 (0.6678) | -0.143 (0.2658) | 0.312 (0.5937)
  Day 4: 72 hours post-dose | 0.290 (1.3130) | 3.907 (6.9842) | -0.107 (0.5805) | 0.257 (1.7737) | 1.617 (0.8663) | -0.423 (0.3927) | 0.163 (0.2829) | -0.282 (0.7349) | -0.327 (9.5142) | -0.383 (0.9286) | 0.473 (0.9347) | 0.398 (1.5906)
  Day 5: 96 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 3 | 6
  Day 5: 96 hours post-dose |  |  |  |  |  |  |  |  | 10.166 (15.4306) | -0.452 (0.7897) | -0.293 (0.6240) | -0.307 (0.4571)
  Day 8: 168 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 3 | 16
  Day 8: 168 hours post-dose | 3.230 (6.0836) | -1.280 (1.1086) | -0.323 (0.7149) | -0.667 (0.7332) | 0.330 (0.1015) | -0.643 (0.0153) | 0.027 (0.0462) | 0.217 (0.3525) | 13.542 (20.3702) | -0.284 (0.4548) | -0.150 (0.6874) | 0.001 (1.7010)
  Day 15: 336 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1 | 2 | 2 | 6 | 5 | 4 | 3 | 15
  Day 15: 336 hours post-dose | 2.023 (1.8553) | 2.310 (4.7039) | -0.287 (0.7174) | -0.067 (1.1829) | 0.930 (NA) — Standard deviaiton is not calculable for 1 value. | -0.550 (0.1273) | 0.000 (0.0000) | 2.898 (7.8222) | -11.698 (14.0227) | -0.703 (1.9050) | 0.257 (1.0000) | 0.081 (1.1008)
  Day 36: 840 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 2 | 2 | 6 | 5 | 5 | 3 | 14
  Day 36: 840 hours post-dose | 2.077 (1.8309) | -1.083 (1.1453) | -0.113 (0.2747) | -0.657 (1.7796) |  | -0.660 (0.0283) | -0.085 (0.1202) | 2.277 (6.9301) | -10.962 (14.6454) | -0.456 (0.8780) | -0.283 (0.5346) | 0.464 (1.5409)
  Day 71: 1680 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 6 | 5 | 3 | 8
  Day 71: 1680 hours post-dose |  |  |  |  |  |  | 0.580 (1.1549) | 10.358 (18.0554) | -9.218 (13.7046) | 0.080 (1.3326) | -0.310 (0.5112) | 1.984 (4.3754)

29. Secondary Outcome: Change From Baseline in Activated Factor B (Bb) at Scheduled Timepoints
Description: Bb was one of the complement components/biomarkers explored in the study. Baseline was defined as the average of measurement on Day -1 and pre-dose (0 hours) measurement on Day 1.
Time Frame: as for outcome 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3 | 16
milligrams per liter (mg/L)
  Day 1: 1 hour post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 1 | 0 | 0 | 10
  Day 1: 1 hour post-dose | 0.277 (0.2574) | 0.177 (0.1106) | 0.680 (0.1735) | 1.897 (1.4677) | 3.713 (1.2371) | 4.130 (0.4888) | -0.073 (0.1563) | -0.518 (1.1527) | 0.000 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | 0.132 (0.2589)
  Day 1: 3 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 1 | 0 | 0 | 10
  Day 1: 3 hours post-dose | 0.057 (0.3636) | 0.253 (0.0473) | 0.593 (0.1943) | 0.977 (0.9903) | 3.920 (1.6404) | 2.850 (0.1838) | 0.117 (0.2011) | -0.015 (0.7729) | 0.120 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | 0.175 (0.3925)
  Day 1: 5 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 6 | 6 | 3 | 16
  Day 1: 5 hours post-dose | -0.117 (0.3980) | -0.243 (0.3557) | 0.117 (0.1150) | 0.260 (0.2762) | 2.313 (2.3526) | 1.355 (0.0636) | 0.163 (0.1626) | -0.253 (1.4442) | 0.048 (0.0560) | 1.013 (0.8021) | 0.673 (0.5974) | 0.031 (0.2548)
  Day 1: 8 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 1 | 0 | 0 | 5
  Day 1: 8 hours post-dose |  |  |  |  | 1.670 (NA) — Standard deviaiton is not calculable for 1 value. | 0.375 (0.3889) | 0.067 (0.3308) | -0.432 (1.5607) | 0.240 (NA) — Standard deviaiton is not calculable for 1 value. |  |  | 0.030 (0.2307)
  Day 1: 12 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 6 | 6 | 3 | 11
  Day 1: 12 hours post-dose |  |  |  |  | 0.830 (NA) — Standard deviaiton is not calculable for 1 value. | 0.145 (0.2051) | 0.097 (0.5154) | -0.318 (1.8083) | 0.198 (0.1277) | 0.775 (0.5881) | 0.523 (0.5636) | -0.015 (0.2355)
  Day 2: 24 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 6 | 6 | 6 | 3 | 16
  Day 2: 24 hours post-dose | -0.360 (0.1637) | -0.097 (0.3465) | -0.233 (0.4041) | -0.577 (1.0866) | 0.377 (0.5680) | 0.315 (0.4455) | 0.030 (0.5565) | -0.322 (1.6140) | 0.220 (0.2082) | 0.908 (1.2157) | 0.413 (0.3602) | -0.016 (0.4309)
  Day 3: 48 hours post-dose | -0.273 (0.0802) | -0.230 (0.3974) | 0.023 (0.0252) | -0.617 (1.1825) | 0.257 (0.4532) | 0.320 (0.5632) | 0.127 (0.6966) | 0.090 (1.5773) | 0.255 (0.2673) | 0.312 (0.5293) | 0.203 (0.2050) | 0.156 (0.7536)
  Day 4: 72 hours post-dose | -0.133 (0.3057) | 0.437 (0.2318) | -0.127 (0.2194) | -0.640 (1.1521) | 0.153 (0.8702) | 0.100 (0.3219) | 0.100 (0.3260) | 0.082 (0.4979) | 0.335 (0.2649) | 0.250 (0.3824) | 0.160 (0.1600) | 0.196 (0.5920)
  Day 5: 96 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 3 | 6
  Day 5: 96 hours post-dose |  |  |  |  |  |  |  |  | 0.372 (0.4206) | -0.016 (0.5003) | 0.053 (0.0462) | -0.018 (0.7665)
  Day 8: 168 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 3 | 16
  Day 8: 168 hours post-dose | -0.423 (0.0961) | -0.217 (0.3121) | -0.067 (0.1155) | -0.657 (1.0185) | 0.110 (0.3772) | 0.083 (0.2940) | -0.050 (0.2787) | -0.047 (0.7904) | 0.158 (0.3306) | -0.522 (0.5220) | 0.057 (0.0981) | 0.187 (0.5747)
  Day 15: 336 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1 | 2 | 2 | 6 | 5 | 4 | 3 | 15
  Day 15: 336 hours post-dose | -0.020 (0.5429) | -0.100 (0.4911) | -0.157 (0.2714) | -0.820 (1.3516) | -0.280 (NA) — Standard deviaiton is not calculable for 1 value. | -0.025 (0.0354) | -0.090 (0.0707) | -0.377 (1.4630) | 0.126 (0.2881) | -0.445 (0.6457) | 0.583 (1.0104) | 0.137 (0.4811)
  Day 36: 840 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 2 | 2 | 6 | 5 | 5 | 3 | 14
  Day 36: 840 hours post-dose | -0.250 (0.2951) | -0.387 (0.4382) | -0.107 (0.3235) | -0.700 (1.0522) |  | 0.360 (0.4525) | 0.450 (0.9617) | -1.018 (1.6763) | 0.890 (1.0579) | -0.040 (0.2539) | 0.163 (0.2329) | 0.266 (0.4960)
  Day 71: 1680 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 6 | 5 | 3 | 8
  Day 71: 1680 hours post-dose |  |  |  |  |  |  | 2.067 (2.8386) | -1.165 (2.2748) | 0.818 (0.5851) | -0.466 (0.4039) | 0.193 (0.3349) | 0.058 (0.5159)

ADVERSE EVENTS:
Time Frame: Baseline (Study Day -2) through study completion (Study Day 36 for IV treatment cohorts, and Study Day 71 SC treatment cohorts).
Description: The time period for actively eliciting and collecting AEs and SAEs ("active collection period") for each participant beginned from the time the participant provides informed consent, which was obtained before the participants participation in the study (ie, before undergoing any study related procedure and/or receiving investigational product), through and including a minimum of 28 calendar days, after the last administration of the investigational product.
Arm/Group | Cohort 1: PF-06755347 0.01 mg/kg IV | Cohort 2: PF-06755347 0.03 mg/kg IV | Cohort 3: PF-06755347 0.1 mg/kg IV | Cohort 4: PF-06755347 0.3 mg/kg IV | Cohort 5: PF-06755347 1 mg/kg IV | Cohort 6: PF-06755347 0.7 mg/kg IV | Cohort 7: PF-06755347 25 mg SC | Cohort 8: PF-06755347 50 mg SC | Cohort 9: PF-06755347 100 mg SC | Cohort 10: PF-06755347 200 mg SC | Cohort 11: PF-06755347 300 mg SC | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/3 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 1/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/3 | 0/16
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 3/3 | 3/3 | 3/3 | 2/3 | 3/3 | 6/6 | 6/6 | 5/6 | 3/3 | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-06755347 0.01 mg/kg IV (N=3) | Cohort 2: PF-06755347 0.03 mg/kg IV (N=3) | Cohort 3: PF-06755347 0.1 mg/kg IV (N=3) | Cohort 4: PF-06755347 0.3 mg/kg IV (N=3) | Cohort 5: PF-06755347 1 mg/kg IV (N=3) | Cohort 6: PF-06755347 0.7 mg/kg IV (N=3) | Cohort 7: PF-06755347 25 mg SC (N=3) | Cohort 8: PF-06755347 50 mg SC (N=6) | Cohort 9: PF-06755347 100 mg SC (N=6) | Cohort 10: PF-06755347 200 mg SC (N=6) | Cohort 11: PF-06755347 300 mg SC (N=3) | Placebo (N=16)
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-06755347 0.01 mg/kg IV (N=3) | Cohort 2: PF-06755347 0.03 mg/kg IV (N=3) | Cohort 3: PF-06755347 0.1 mg/kg IV (N=3) | Cohort 4: PF-06755347 0.3 mg/kg IV (N=3) | Cohort 5: PF-06755347 1 mg/kg IV (N=3) | Cohort 6: PF-06755347 0.7 mg/kg IV (N=3) | Cohort 7: PF-06755347 25 mg SC (N=3) | Cohort 8: PF-06755347 50 mg SC (N=6) | Cohort 9: PF-06755347 100 mg SC (N=6) | Cohort 10: PF-06755347 200 mg SC (N=6) | Cohort 11: PF-06755347 300 mg SC (N=3) | Placebo (N=16)
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Administration site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Application site irritation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 3
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 2 | 2 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram PR prolongation (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Penile erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perineal swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to sponsor's business decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT03275740/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT03275740/SAP_001.pdf